CLINICAL TRIAL: NCT04489173
Title: A Phase 2 Study of Trifluridine/Tipiracil in Patients With ER-positive, HER2-negative Advanced Breast Cancer That Previously Received Chemotherapy
Brief Title: TAS102 in Patients With ER-positive, HER2-negative Advanced Breast Cancer
Acronym: TIBET
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Borstkanker Onderzoek Groep (Network)
Collaborators: Erasmus Medical Center (Other); UMC Utrecht (Other); Servier (Industry); BOOG Study Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BOOG 2019-01
Record Dates: First submitted 2020-07-22; First posted 2020-07-28 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Breast Neoplasm; Chemotherapy Effect
Keywords: TAS102
MeSH Terms: conditions — Breast Neoplasms | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Intervention Model Description: Multicenter, single arm, phase 2 study evaluating the efficacy and safety of trifluridine/tipiracil in women with metastatic or locally advanced breast cancer not amenable to curative treatment by surgery or radiotherapy.
  Study medication should be started within 3 days after completion of screening and continue until a study treatment discontinuation criterion is met.
  Trifluridine/tipiracil will be administered orally BID on days 1 through 5, with the first dose administered in the morning of day 1 of each cycle and the last dose administered in the evening of day 5, followed by a recovery period from day 6 through day 7. Trifluridine/tipiracil will be administered orally BID on days 8 through 12, with the first dose administered in the morning of day 8 of each cycle and the last dose administered in the evening of day 12, followed by a recovery period from day 13 through day 28. Each cycle will be 28 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Treatment with TAS102
  Interventions: Drug: trifluridine/tipiracil

INTERVENTIONS:
Drug: trifluridine/tipiracil — Study medication should be started within 3 days after completion of screening and continue until a study treatment discontinuation criterion is met.
  Trifluridine/tipiracil will be administered orally BID on days 1 through 5, with the first dose administered in the morning of day 1 of each cycle and the last dose administered in the evening of day 5, followed by a recovery period from day 6 through day 7. Trifluridine/tipiracil will be administered orally BID on days 8 through 12, with the first dose administered in the morning of day 8 of each cycle and the last dose administered in the evening of day 12, followed by a recovery period from day 13 through day 28. Each cycle will be 28 days.
  Other Names: Lonsurf, TAS102

SUMMARY:
This is a multicenter phase 2 study evaluating the efficacy and safety of trifluridine/tipiracil in women with metastatic or locally advanced breast cancer not amenable to curative treatment by surgery or radiotherapy.

DETAILED DESCRIPTION:
Multicenter phase 2 study evaluating the efficacy and safety of trifluridine/tipiracil in women with metastatic or locally advanced breast cancer not amenable to curative treatment by surgery or radiotherapy. This study will be conducted under the sponsorship of BOOG, Amsterdam, NL.

Objectives:

To evaluate the efficacy of trifluridine/tipiracil by determination of the percentage of patients being progression free at 8 weeks on trifluridine/tipiracil prescribed for ER-positive, HER2-negative advanced breast cancer patients previously treated with a taxane and capecitabine.

Endpoints:

Progression-free survival at 8 weeks.

Progression-free survival.

Response rate CR/PR at 16 weeks.

Adverse events.

Translational research on biological factors that may be of influence on the outcome of treatment.

QoL.

Main eligibility criteria:

Metastatic Her2 negative, ER-positive breast cancer patients that progressed on, or after treatment with Capecitabine. Previous treatment with Taxanes is obligatory. Adequate hematology, liver and renal function tests.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women(≥ 18 years of age) with proven diagnosis of metastatic or locally advanced breast cancer not amenable to curative treatment by surgery or radiotherapy
2. Documented ER positive (10%) and/or PR positive (10%) and HER2 negative metastatic breast cancer
3. Progressive disease based on imaging
4. Women previously treated with capecitabine (in metastatic setting), and a maximum of two other lines of chemotherapy including a taxane either in the (neo)adjuvant or metastatic setting.
5. Evaluable disease as defined per RECIST v.1.1 (see Appendix B). Tumor lesions previously irradiated or subjected to other locoregional therapy will only be deemed measurable if disease progression at the treated site after completion of therapy is clearly documented.
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
7. Life expectancy of ≥ 12 weeks
8. Willing and able to comply with scheduled visits and study procedures
9. Adequate organ, bone marrow and coagulation function as shown by:

   * Absolute neutrophil count (ANC) ≥ 1.5 ×109/L
   * Platelets ≥ 75 ×109/L
   * Hemoglobin (Hgb) ≥ 5.6 mmol/L
   * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 ULN (or ≤ 5 if hepatic metastases are present)
   * Total serum bilirubin ≤ 1.5 × ULN (≤ 3 × ULN for patients known to have Gilbert Syndrome)
   * Creatinine clearance ≥60 ml/min
10. Written informed consent obtained before any screening procedure and according to local guidelines.
11. Resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to NCI CTCAE version 4.0 Grade ≤1, except alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion.

Exclusion Criteria:

1. HER2-overexpressing patients by local laboratory testing (IHC 3+ staining or in situ hybridization positive) and ER-negative patients are not eligible
2. No more than two lines of chemotherapy for advanced disease
3. Resolution of side-effects from previous chemotherapy > grade 1 (except for alopecia)
4. Radiotherapy within four weeks prior to enrollment is not allowed except in case of localized radiotherapy for analgesic purpose or for lytic lesions at risk of fracture which can then be completed within two weeks prior to enrollment. Patients must have recovered from radiotherapy toxicities prior to enrollment.
5. 30% or more marrow-bearing bone being irradiated. Other primary tumors within the last 5 years before study entry are not allowed, except for adequately controlled basal cell carcinoma of the skin, or carcinoma in situ of the cervix.
6. Previous or current CNS metastases, carcinomatous meningitis, are not allowed. A CT or MRI of the brain must be performed within 4 weeks prior to registration if the presence of metastases at this site is suspected.
7. Evidence of clinically significant cardiovascular or pulmonary disease or any other disease, metabolic or psychological dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, or that may affect patient compliance with study routines, or places the patient at high risk from treatment related complications. (e.g lactose intolerance)
8. Previously received trifluridine/tipiracil
9. Since trifluridine/tipiracil contains lactose, patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption should not take this medicine
10. Diagnosis of any other malignancy prior to registration, except those that are not believed to influence the patient's prognosis and do not require any further treatment.
11. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 8 weeks
  Response rate CR/PR

SECONDARY OUTCOMES:
Adverse events | every 4 weeks
  CTCAE version 4.0
QoL | 32 weeks
  Quality of Life questionnaire EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: A. Elise van Leeuwen-Stok, PhD, Study Director — BOOG Study Center
Locations (10):
- Netherlands (10):
  - Rijnstate, Arnhem
  - Wilhelmina ziekenhuis, Assen
  - Amphia Ziekenhuis, Breda
  - Reinier de Graaf Groep, Delft
  - Deventer ziekenhuis, Deventer
  - Catharina Ziekenhuis, Eindhoven
  - MC Leeuwarden, Leeuwarden
  - MUMC, Maastricht
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guchelaar NAD, Mathijssen RHJ, de Boer M, van Bekkum ML, Heijns JB, Vriens BEPJ, van Rosmalen MM, Kessels LW, Hamming L, Beelen KJ, Nieboer P, van den Berg SM, Hoop EO, Bijlsma RM, Bos MEMM; Dutch Breast Cancer Research Group (BOOG). Trifluridine-tipiracil in previously treated patients with oestrogen receptor-positive, HER2-negative metastatic breast cancer (BOOG 2019-01 TIBET trial): a single-arm, multicentre, phase 2 trial. EClinicalMedicine. 2025 Jan 27;80:103065. doi: 10.1016/j.eclinm.2024.103065. eCollection 2025 Feb. PMID 40017682